CLINICAL TRIAL: NCT04959591
Title: Use of Intravenous Acetaminophen in Adolescents and Pediatrics Undergoing Spinal Fusion Surgery: Randomized Controlled Trial
Brief Title: Use of Intravenous Acetaminophen in Pediatrics Undergoing Spinal Fusion Surgery
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Asan Medical Center (Other)
Responsible Party: Principal Investigator, Won Uk, Koh, Associate professor, Asan Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2021-0411
Record Dates: First submitted 2021-06-28; First posted 2021-07-13 (Actual); Last update posted 2022-12-28 (Actual); Status verified 2022-12

CONDITIONS: Scoliosis; Adolescence
Keywords: scoliosis, acetaminophen
MeSH Terms: conditions — Scoliosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The designated research pharmacist will prepare the both study drug (IV acetaminophen) and placebo and will dispense the study drug according to treatment allocation. Treatment allocation will remain concealed from all other investigators involved in the conduct and analysis of the trial. All other medical staff involved in patient care during the hospital stay of study participant and the study participants itself along with guardians will be also blinded throughout.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Experimental (Pre): Acetaminophen (Experimental): Participants will receive 15mg/kg intravenous acetaminophen 15mg/kg after anesthetic induction/before surgical incision and the same dose will be given postoperatively at 8 hour intervals for 24hours. A single dose of placebo (saline) will also be given at the end of surgery before skin closure.
  Interventions: Drug: intravenous acetaminophen
- Experimental(post): Acetaminophen (Experimental): Participants will receive 15mg/kg intravenous acetaminophen 15mg/kg at the end of surgery before skin closure and the same dose will be given postoperatively at 8 hour intervals for 24hours. A single dose of placebo (saline) will also be given after anesthetic induction/before surgical incision.
  Interventions: Drug: intravenous acetaminophen
- Placebo comparator : placebo (Placebo Comparator): Participants will receive 1.5ml/kg placebo (0.9% saline) before and after surgery and the same dose will be given postoperatively at 8hour intervals for 24hours.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: intravenous acetaminophen — experimental(pre): administration of IV acetaminophen
  Arms: Experimental (Pre): Acetaminophen
Drug: intravenous acetaminophen — experimental(post): administration of IV acetaminophen
  Arms: Experimental(post): Acetaminophen
Drug: Placebo — placebo comparator: administration of normal saline
  Arms: Placebo comparator : placebo

SUMMARY:
The purpose of this study is to investigate whether perioperative intravenous acetaminophen administration reduces postoperative pain and opioid consumption in adolescents and pediatric patients undergoing spinal fusion surgery.

DETAILED DESCRIPTION:
Spinal fusion surgery to correct scoliosis causes severe postoperative pain in adolescents and pediatric patients. Thus, appropriate control of postoperative pain has a significant impact on postoperative recovery, patient satisfaction and reduction of hospital stay. Although pain control was achieved through only opioids, the importance of multimodal analgesia has recently been emphasized as opioid addiction and side effects increase.

Acetaminophen is recommended as a key factor in multimodal analgesia and previous studies performed in adult spine surgery showed that intravenous administration of acetaminophen reduced the postoperative pain and opioid consumption. In addition, acetaminophen is a drug widely recognized for safety in adolescents and pediatric patients and has a fast and predictable analgesic effect. Therefore, the purpose of this study is to investigate whether perioperative intravenous acetaminophen administration reduces postoperative pain and opioid consumption in adolescents and pediatric patients undergoing spinal fusion surgery. Thus the specific aim of this trial the investigators will determine is;

1. The decrease in postoperative analgesic requirement following IV acetaminophen
2. The decrease in intensity of postoperative pain following IV acetaminophen
3. The quality of recovery including self-reported recovery, physical and functional recovery and length of stay
4. The preemptive analgesic effect of IV acetaminophen

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) physical status 1-3
* patients undergoing spinal fusion surgery

Exclusion Criteria:

* patients who refuse to participate in this study
* patients unable to communicate due to mental impairment or developmental delay
* patients allergic to acetaminophen or its additives or who are contraindicated in acetaminophen administration for other reasons
* patients with existing liver diseases or dysfunction (i.e. active hepatitis, clinically relevant chronic liver conditions, elevated liver enzymes)
* patients who are judged ineligible by the medical staff to participate in the study for other reasons

Ages: 11 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 99 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2022-04-15 (Actual); Study Completion 2022-04-22 (Actual)

PRIMARY OUTCOMES:
Postoperative analgesic consumption | 24 hours after surgery
  Comparison of total analgesic consumption between 3 groups in morphine equivalent

SECONDARY OUTCOMES:
Postoperative analgesic consumption | 48 hours after surgery
  Comparison of total analgesic consumption between 3 groups in morphine equivalent
Post operative pain scores | 4, 8, 24, 48 hours after surgery
  Comparison of NRS(numerical rating scale: 0, no pain, 10, worst possible pain) between 3 groups: Worst (cough) and mean pain scores
Frequency of side effects of opioids | 24, 48, 72 hours after surgery
  respiratory depression, postoperative nausea/vomiting, itching, constipation
Quality of recovery questionaire | 3 to 5 days after surgery
  self reported Quality of recovery-15 (QoR-15: 0, very poor recovery, 150, excellent recovery) questionnaire
Postoperative recovery | from end of surgery to discharge from hospitalization (average 7 days)
  Timing of oral intake(hr), timing of ambulation(hr)
Length of hospital day | from end of surgery to discharge from hospitalization (average 7 days)
  postoperative hospital stay(days), intensive care unit admission(days)

CONTACTS AND LOCATIONS:
Overall Officials: Won Uk Koh, M.D, Ph.D, Principal Investigator — Asan Medical Center
Locations (1):
- Asan Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Shastri N. Intravenous acetaminophen use in pediatrics. Pediatr Emerg Care. 2015 Jun;31(6):444-8; quiz 449-50. doi: 10.1097/PEC.0000000000000463. PMID 26035501
- [Background] Wick EC, Grant MC, Wu CL. Postoperative Multimodal Analgesia Pain Management With Nonopioid Analgesics and Techniques: A Review. JAMA Surg. 2017 Jul 1;152(7):691-697. doi: 10.1001/jamasurg.2017.0898. PMID 28564673
- [Background] Ceelie I, de Wildt SN, van Dijk M, van den Berg MM, van den Bosch GE, Duivenvoorden HJ, de Leeuw TG, Mathot R, Knibbe CA, Tibboel D. Effect of intravenous paracetamol on postoperative morphine requirements in neonates and infants undergoing major noncardiac surgery: a randomized controlled trial. JAMA. 2013 Jan 9;309(2):149-54. doi: 10.1001/jama.2012.148050. PMID 23299606
- [Derived] Kim YJ, Kim HJ, Kim S, Kim H, Lee CS, Hwang CJ, Cho JH, Ro YJ, Koh WU. Comparison of preemptive and preventive intravenous acetaminophen on opioid consumption in pediatrics undergoing posterior spinal fusion surgery: a randomized controlled trial. Korean J Anesthesiol. 2024 Jun;77(3):326-334. doi: 10.4097/kja.23747. Epub 2024 Feb 20. PMID 38383005